CLINICAL TRIAL: NCT03706495
Title: The Effect of Functional Exercises on Balance With Postural Thoracic Kyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, sena ozdemir, Assistant Prof., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10840098-604.01.01
Record Dates: First submitted 2018-09-04; First posted 2018-10-16 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Postural Kyphosis; Balance
Keywords: Postural Kyphosis; Exercises; Balance; Respiratory Functions
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized double-blind
Who Masked: Participant, Investigator
Masking Description: Participants involved in the study and the physiotherapist doing the assessment do not know which exercise group they will be involved in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Group I (Experimental): The Group I Postural exercise will receive postural exercise for 60 min/day 2 times/week for 8 weeks.
  Interventions: Behavioral: The Group I Postural Exercise
- The Group II (Experimental): The Schroth method three-dimensional exercise therapy program consists of individual exercise programs combined with correction patterns. It is based on sensorimotor and kinesthetic principles. Goals of this exercise are to facilitate the correction of the asymmetric posture and to maintain the correct posture in the daily activities of the patient. The Group II receive Schroth method based on three-dimensional exercise therapy program for 60 min/day 2 times/week for 8 weeks.
  Interventions: Behavioral: The Group II Three-dimensional Exercise Therapy Program

INTERVENTIONS:
Behavioral: The Group I Postural Exercise — Spine anatomy and daily life activities will be informed about proper posture. Strengthening of postural muscles, stretching (Pectoral Region, M. Psoas Major) and breathing exercise will be performed under the supervision of a physiotherapist. The Group I will receive postural exercise for 60 min/day 2 times/week for 8 weeks.
  Other Names: The Group I Postural Exercise Program
  Arms: The Group I
Behavioral: The Group II Three-dimensional Exercise Therapy Program — The Group II Schroth method corrects the kyphotic posture, with the help of proprioceptive and exteroceptive stimulation and mirror control in the sagittal plane, using specific corrective breathing patterns. The Schroth method three-dimensional exercise therapy program adapted for the specific posture will be exercised in four specific positions (sitting, supine, standing, prone) under the supervision of a physiotherapist. Exercise include, trunk elongation, symmetrical sagittal straightening, shoulder traction, corrective breathing and muscle activation by increasing tension (isometric tension). The Group II will receive Schroth's three-dimensional exercise therapy program for 60 min/day 2 times/week for 8 weeks.
  Other Names: The Group II Schroth Exercise Therapy Program
  Arms: The Group II

SUMMARY:
In a normal spine, the sagittal plane has four curvatures that balance each other. The cervical and lumbar spine is lordotic, the thoracic spine and sacral region are kyphotic. In the sagittal plane, there is an average of 40 kyphosis angles between the T1 vertebrae upper end plate and the T12 vertebra lower end plate. Thoracic kyphosis is defined as an increase in the normal thoracic curvature (above 40) of the spine. Postural kyphosis usually occurs when individuals with weak muscle strength exert excessive external loads on their vertebrae. In rapidly growing young people, the abnormal flexion of the spine prevents the development of internal organs and excess thoracic kyphosis causes changes in respiratory functions, as well as postural disorders negatively affect the standing balance. In addition, the posture and appearance of young people with postural kyphosis are affected, which can affect their physical and psychological health.The incidence of hyper-kyphosis abnormality was reported to be 15.3% in 11 year-old children, 38% in 20 to 50 years old adults and 35% in 20 to 64 years old adults. This abnormality is managed by various methods including manual therapy, postural retraining, taping, orthoses and corrective exercises.

When a literature review was conducted, it was observed that no balance evaluation was performed in individuals between 18 and 25 years of age who had postural kyphosis. Therefore, the aim of this study was to investigate the effect of Schroth-based functional exercise and postural exercise on balance, respiratory functions and thoracic angle, who has with postural kyphosis and 18-25 years of age.

DETAILED DESCRIPTION:
Participants will be randomly allocate 40 participants with kyphosis to two groups; Group I (n=20), Group II (n=20). The Group I, will receive postural exercise for 60 min/day 2 times/week for 8 weeks, while the Group II receive Schroth three-dimensional exercise therapy program for 60 min/day 2 times/week for 8 weeks. Assessment procedure will be held at the beginning and 9th week of study. All subjects will be assessed by each angle of thoracic kyphosis, forward head and forward shoulder angles were measured by using the lateral photographic method, trunk flexibility (lateral and hyperextension), balance (BİODEX balance system) , respiratory function test (measurement of pulmonary function and respiratory muscle strength) , Quality of life SRS-22 and Numeric Rating Scale for pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 25 years,
* Thoracic kyphosis angle ≥ 40,
* Not being treated for kyphosis within the last six months.

Exclusion Criteria:

* Who has mental problem,
* Spinal fractures and / or operative stories,
* Shoulder joint injury,
* Participants who can not come to the exercise program.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Angle of thoracic kyphosis | Baseline
  Spinal alignment was evaluated using a Spinal Mouse (ValedoShape-Hocoma), a computer-assisted noninvasive device. The method has no medical risk or danger. The spinal processes of the vertebra from C7 to S3 were marked. The Spinal Mouse device was slid along the spine from top to bottom to complete the measurement. The evaluation was administered while the subjects were standing in upright position.

SECONDARY OUTCOMES:
Balance Assessment (postural stability test) | Baseline and 9 weeks
  BIODEX balance systems use any of four test protocols including fall risk, athletic single leg stability, limits of stability and postural stability. With the Biodex Balance System, the balance of all participants will be evaluated by postural stability test. The Postural Stability test emphasizes a patient's ability to maintain a center of balance. The patient's score, or "Stability Index", on this test assesses deviations from center, thus a lower score is more desirable than a higher score.
Numeric Rating Scale for Pain | Baseline and 9 weeks
  The Numeric Rating Scale (NRS) for pain is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. The common format is a horizontal bar or line. The pain NRS is a single 11-point numeric scale, an 11-point numeric scale (NRS 11) with 0 representing one pain extreme ("no pain") and 10 representing the other pain extreme ("pain as bad as you can imagine" and "worst pain imaginable").The NRS will be used for pain assessment of the thoracic region.
Forward head and forward shoulder angles | Baseline and 9 weeks
  The lateral photogrammetric measurement method was used to measure the angle of the head protrusion in the tragus-C7 and the proximal C7-acromion in the shoulders.
Trunk Flexibility Assesment | Baseline and 9 weeks
  To asses trunk flexibility, the body will be used for measurement of hyperextension and lateral flexion.
Measurement of pulmonary function | Baseline and 9 weeks
  The desktop spirometer (Cosmed-Pony FX®) is a hand-held instrument for assessment, will be used for pulmonary function test including forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and ratio of FEV1/FVC. Pulmonary function will test following the guidelines recommended by the American Thoracic Society (ATS).Participant, sitting in an upright position comfortably on a chair with nose clip attached and head slightly elevated. They will perform each test for three trials. The best value of each parameter will record. The values express as both an absolute value in liters and a percentage of the predicted normal value.
Measurement of respiratory muscle strength | Baseline and 9 weeks
  The desktop spirometer (Cosmed-Pony FX®) is a hand-held instrument for assessment respiratory muscles strength both inspiratory and expiratory muscles. Inspiratory and expiratory muscles strength is expressed in term of Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP), respectively. MIP and MEP are readily and digitally monitored in units of cmH2O ( pressure range ± 200 cmH2O).
Quality of Life Questionnaire | Baseline and 9 weeks
  The Scoliosis Research Society-22 (SRS-22) questionnaire will be used to assess the quality of life. Turkish validity and reliability studies were conducted. It consists of 22 questions with five subgroups. These subgroups are; pain, image / appearance, function / activity, mental health and treatment satisfaction. For each question, 1 (worst) and 5 (best) were defined as points.

CONTACTS AND LOCATIONS:
Overall Officials: Candan Algun, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seidi F, Rajabi R, Ebrahimi I, Alizadeh MH, Minoonejad H. The efficiency of corrective exercise interventions on thoracic hyper-kyphosis angle. J Back Musculoskelet Rehabil. 2014;27(1):7-16. doi: 10.3233/BMR-130411. PMID 23948845
- [Background] Feng Q, Wang M, Zhang Y, Zhou Y. The effect of a corrective functional exercise program on postural thoracic kyphosis in teenagers: a randomized controlled trial. Clin Rehabil. 2018 Jan;32(1):48-56. doi: 10.1177/0269215517714591. Epub 2017 Jun 14. PMID 28610442
- [Background] Berdishevsky H. Outcome of intensive outpatient rehabilitation and bracing in an adult patient with Scheuermann's disease evaluated by radiologic imaging-a case report. Scoliosis Spinal Disord. 2016 Oct 14;11(Suppl 2):40. doi: 10.1186/s13013-016-0094-7. eCollection 2016. PMID 27785478
- [Background] Singla D, Veqar Z. Association Between Forward Head, Rounded Shoulders, and Increased Thoracic Kyphosis: A Review of the Literature. J Chiropr Med. 2017 Sep;16(3):220-229. doi: 10.1016/j.jcm.2017.03.004. Epub 2017 Sep 28. PMID 29097952
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Derived] Ozdemir Gorgu S, Algun ZC. A randomized controlled study of the effect of functional exercises on postural kyphosis: Schroth-based three-dimensional exercises versus postural corrective exercises. Disabil Rehabil. 2023 Jun;45(12):1992-2002. doi: 10.1080/09638288.2022.2083244. Epub 2022 Jun 12. PMID 35694970